CLINICAL TRIAL: NCT06342362
Title: Neuroprotective Outcomes of Magnesium Sulfate in Neonates With Hypoxic-Ischemic Encephalopathy (HIE) at Tertiary Care Hospital of Karachi
Brief Title: Magnesium Sulfate in Neonatal HIE"
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sindh Institute of Child Health and Neonatology (Other)
Responsible Party: Principal Investigator, Sher Wali Khan, fellow Neonatologist, Sindh Institute of Child Health and Neonatology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SICHN/IRB-001/2024
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Neonates With HIE
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (receiving magnesium sulfate) (Experimental): Participants would be randomly assigned to either the treatment group (receiving magnesium sulfate) or the control group (receiving a placebo or standard treatment).
  Interventions: Drug: Magnesium sulfate
- the control group (receiving a placebo or standard treatment) (Placebo Comparator): Participants would be randomly assigned to either the treatment group (receiving
  Interventions: Other: placebo or standard treatment)

INTERVENTIONS:
Drug: Magnesium sulfate — Participants would be randomly assigned to either the treatment group (receiving magnesium sulfate) or the control group (receiving a placebo or standard treatment).
  Arms: treatment group (receiving magnesium sulfate)
Other: placebo or standard treatment) — placebo or standard treatment)
  Arms: the control group (receiving a placebo or standard treatment)

SUMMARY:
The study will investigates the neuroprotective effects of intravenous magnesium sulfate in neonates with hypoxic-ischemic encephalopathy (HIE) at a Karachi tertiary care hospital. Using a randomized clinical trial design, the study targets term and near-term newborns with moderate to severe HIE. Data collection involves obtaining informed consent, preparing and administering magnesium sulfate, and assessing outcomes including mortality and morbidity. The study aims to provide insights into improving patient outcomes and clinical practice for neonatal HIE management.

DETAILED DESCRIPTION:
Objective:

• To determine the neuroprotective outcomes of intravenous magnesium sulphate in neonates with hypoxic ischemic encephalopathy (HIE) at a tertiary care hospital of Karachi.

Methodology:

* Study Setting: This is a prospective study; and will be conducted at tertiary care hospital of Karachi (Sindh Institute of Child Health and Neonatology, K-5).
* Study Design: Rndomized clinical Trial
* Target Population: The study population will be all term and near term newborns (≥35 completed weeks) with moderate to severe HIE.
* Inclusion Criteria: All Late preterm and term newborn with hypoxic ischemic encephalopathy (HIE) on basis of sarnat score and reaching in our unit within 6 hours of life will be the part of our trial.
* Exclusion Criteria:

  * Newborns of less than 34 weeks, with dimorphism, comorbidities or arriving after 6 hours of birth, will be excluded.
  * Pre-existing medical conditions that may interfere with the assessment of neuroprotective outcomes.
  * Congenital anomalies or genetic disorders affecting neurological function.
  * Allergy or known adverse reactions to magnesium sulfate.
  * Participation in another concurrent clinical trial involving investigational drugs or interventions.
  * Inability to obtain informed consent from parents or guardians.
* Medical Intervention: Magnesium sulphate as infusion will be commenced to cases. Control will be treated as per unit protocol.

Sample Size:

Sample size was calculated using WHO software with the following assumptions:

Level of significance α=0.05 Power of study = 80 Anticipated population proportion P1 = 0.657 Anticipated population proportion P2 = 0.3757 Desired precision = 5 Required sample size 51 for each population (cases 51 and control 51) so, the total 102 is the minimum sample

ELIGIBILITY:
Inclusion Criteria: All Late preterm and term newborn with hypoxic ischemic encephalopathy (HIE) on basis of sarnat score and reaching in our unit within 6 hours of life will be the part of our trial.

-

Exclusion Criteria:

* Newborns of less than 34 weeks, with dimorphism, comorbidities or arriving after 6 hours of birth, will be excluded.
* Pre-existing medical conditions that may interfere with the assessment of neuroprotective outcomes.
* Congenital anomalies or genetic disorders affecting neurological function.
* Allergy or known adverse reactions to magnesium sulfate.
* Participation in another concurrent clinical trial involving investigational drugs or interventions.
* Inability to obtain informed consent from parents or guardians.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2024-04-02 (Estimated); Primary Completion 2024-10-02 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
Neuroprotective effects | 6 months
  Neuroprotective effects: decrease in the frequency or duration of seizures, ability to suck

CONTACTS AND LOCATIONS:
Locations (1):
- SICHN, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No